CLINICAL TRIAL: NCT04687709
Title: To Investigate the Role of Gut Microbiome in Androgen Deprivation Therapy Related Metabolic Changes in Prostate Cancer Patients
Brief Title: To Investigate the Role of Gut Microbiome in ADT Related Metabolic Changes in Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2020.603
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Total bacterial DNA will be extracted from fecal samples by using the bead-beating method with Qiagen QIAamp PowerFecal Pro DNA kit. The extracted DNA will be quantified by Nanodrop for polymerase chain reaction (PCR)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate cancer is the second most common cancer in male cancer globally and ranked third in Hong Kong. While androgen deprivation therapy (ADT) is the backbone treatment for advanced prostate cancer, it could lead to obesity, metabolic syndrome and increased cardiovascular mortality. Previous studies showed that ADT patients have different gut microbiome compared to non-ADT patients and the gut microbiome might be related to the metabolic changes. However, the underlying mechanism of these metabolic complications is still not fully understood. This study aims to investigate the relationship and related mechanism between the changes in gut microbiomes and ADT-related metabolic change in prostate cancer patients.

DETAILED DESCRIPTION:
It is a prospective longitudinal observational human study. Fifty prostate cancer patients planned for ADT will be recruited. Fecal sample will be collected before initiation of ADT, and then at 3 and 6 months after initiation of ADT. Anthropometric, blood metabolic parameters, serum inflammation markers and panels of microbiome metabolites will be measured at these timepoints. Changes in gut microbiome from baseline to 6 months after initiation of ADT will be assessed. Correlation of changes in gut microbiome and metabolic changes, as well as inflammation and microbiome metabolites, will be assessed and possible mechanisms will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject with age 45 or above
2. Histological diagnosis of prostate cancer (acinar type)
3. Clinically decided for androgen deprivation therapy (ADT) as treatment for prostate cancer

Exclusion Criteria:

1. History of diabetes
2. Patients that have other active treatment for prostate cancer or other cancers (except ADT)
3. Patients received treatment, either surgical or medical, that could lead to decrease in serum testosterone prior to commencement of ADT
4. Patients will be started on other treatments, including chemotherapy, new generation of androgen-receptor targeted agents, radiotherapy etc, within 6 months of the commencement of ADT.
5. Subject with recent antibiotics usage within 3 months.

Min Age: 45 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with prostate cancer and is going to receive ADT treatment will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
To assess the changes in gut microbiota in prostate cancer patients after initiation of androgen deprivation therapy (ADT) | Baseline, Month 3, Month 6
  Gut microbiome related metabolites will be measured by ELISA and mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan SY, Ng CF, Lee KW, Yee CH, Chiu PK, Teoh JY, Hou SS. Differences in cancer characteristics of Chinese patients with prostate cancer who present with different symptoms. Hong Kong Med J. 2017 Feb;23(1):6-12. doi: 10.12809/hkmj164875. Epub 2016 Dec 9. PMID 27932742
- [Background] Dao MC, Clement K. Gut microbiota and obesity: Concepts relevant to clinical care. Eur J Intern Med. 2018 Feb;48:18-24. doi: 10.1016/j.ejim.2017.10.005. Epub 2017 Oct 27. PMID 29110901
- [Background] Wong MC, Goggins WB, Wang HH, Fung FD, Leung C, Wong SY, Ng CF, Sung JJ. Global Incidence and Mortality for Prostate Cancer: Analysis of Temporal Patterns and Trends in 36 Countries. Eur Urol. 2016 Nov;70(5):862-874. doi: 10.1016/j.eururo.2016.05.043. Epub 2016 Jun 8. PMID 27289567
- [Background] Saylor PJ, Smith MR. Adverse effects of androgen deprivation therapy: defining the problem and promoting health among men with prostate cancer. J Natl Compr Canc Netw. 2010 Feb;8(2):211-23. doi: 10.6004/jnccn.2010.0014. PMID 20141678
- [Background] Teoh JY, Chan SY, Chiu PK, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of acute myocardial infarction after androgen-deprivation therapy for prostate cancer in a Chinese population. BJU Int. 2015 Sep;116(3):382-7. doi: 10.1111/bju.12967. Epub 2015 Mar 7. PMID 25327618
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of ischemic stroke after androgen deprivation therapy for prostate cancer in the Chinese population living in Hong Kong. Jpn J Clin Oncol. 2015 May;45(5):483-7. doi: 10.1093/jjco/hyv025. Epub 2015 Feb 26. PMID 25724216
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of new-onset diabetes after androgen deprivation therapy for prostate cancer in the Asian population. J Diabetes. 2015 Sep;7(5):672-80. doi: 10.1111/1753-0407.12226. Epub 2014 Dec 22. PMID 25266491
- [Background] Wong SH, Kwong TNY, Wu CY, Yu J. Clinical applications of gut microbiota in cancer biology. Semin Cancer Biol. 2019 Apr;55:28-36. doi: 10.1016/j.semcancer.2018.05.003. Epub 2018 May 18. PMID 29782923
- [Background] Li JKM, Chiu PKF, Ng CF. The impact of microbiome in urological diseases: a systematic review. Int Urol Nephrol. 2019 Oct;51(10):1677-1697. doi: 10.1007/s11255-019-02225-y. Epub 2019 Jul 12. PMID 31301004
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309
- [Background] Dabke K, Hendrick G, Devkota S. The gut microbiome and metabolic syndrome. J Clin Invest. 2019 Oct 1;129(10):4050-4057. doi: 10.1172/JCI129194. PMID 31573550
- [Background] Boutagy NE, McMillan RP, Frisard MI, Hulver MW. Metabolic endotoxemia with obesity: Is it real and is it relevant? Biochimie. 2016 May;124:11-20. doi: 10.1016/j.biochi.2015.06.020. Epub 2015 Jun 29. PMID 26133659
- [Background] den Besten G, van Eunen K, Groen AK, Venema K, Reijngoud DJ, Bakker BM. The role of short-chain fatty acids in the interplay between diet, gut microbiota, and host energy metabolism. J Lipid Res. 2013 Sep;54(9):2325-40. doi: 10.1194/jlr.R036012. Epub 2013 Jul 2. PMID 23821742
- [Background] Neuman H, Debelius JW, Knight R, Koren O. Microbial endocrinology: the interplay between the microbiota and the endocrine system. FEMS Microbiol Rev. 2015 Jul;39(4):509-21. doi: 10.1093/femsre/fuu010. Epub 2015 Feb 19. PMID 25701044
- [Background] Santos-Marcos JA, Rangel-Zuniga OA, Jimenez-Lucena R, Quintana-Navarro GM, Garcia-Carpintero S, Malagon MM, Landa BB, Tena-Sempere M, Perez-Martinez P, Lopez-Miranda J, Perez-Jimenez F, Camargo A. Influence of gender and menopausal status on gut microbiota. Maturitas. 2018 Oct;116:43-53. doi: 10.1016/j.maturitas.2018.07.008. Epub 2018 Jul 19. PMID 30244778
- [Background] Zhao H, Chen J, Li X, Sun Q, Qin P, Wang Q. Compositional and functional features of the female premenopausal and postmenopausal gut microbiota. FEBS Lett. 2019 Sep;593(18):2655-2664. doi: 10.1002/1873-3468.13527. Epub 2019 Jul 17. PMID 31273779
- [Background] Harada N, Hanaoka R, Horiuchi H, Kitakaze T, Mitani T, Inui H, Yamaji R. Castration influences intestinal microflora and induces abdominal obesity in high-fat diet-fed mice. Sci Rep. 2016 Mar 10;6:23001. doi: 10.1038/srep23001. PMID 26961573
- [Background] Gao W, Wu D, Wang Y, Wang Z, Zou C, Dai Y, Ng CF, Teoh JY, Chan FL. Development of a novel and economical agar-based non-adherent three-dimensional culture method for enrichment of cancer stem-like cells. Stem Cell Res Ther. 2018 Sep 26;9(1):243. doi: 10.1186/s13287-018-0987-x. PMID 30257704
- [Background] Tsoi TH, Chan CF, Chan WL, Chiu KF, Wong WT, Ng CF, Wong KL. Urinary Polyamines: A Pilot Study on Their Roles as Prostate Cancer Detection Biomarkers. PLoS One. 2016 Sep 6;11(9):e0162217. doi: 10.1371/journal.pone.0162217. eCollection 2016. PMID 27598335
- [Background] Teoh JY, Ng CF. Cardiovascular risk after androgen deprivation therapy for prostate cancer: an Asian perspective. Int Urol Nephrol. 2016 Sep;48(9):1429-35. doi: 10.1007/s11255-016-1337-5. Epub 2016 Jun 2. PMID 27256399
- [Background] Cheung MK, Lam WY, Fung WY, Law PT, Au CH, Nong W, Kam KM, Kwan HS, Tsui SK. Sputum microbiota in tuberculosis as revealed by 16S rRNA pyrosequencing. PLoS One. 2013;8(1):e54574. doi: 10.1371/journal.pone.0054574. Epub 2013 Jan 24. PMID 23365674
- [Background] Hui AW, Lau HW, Chan TH, Tsui SK. The human microbiota: a new direction in the investigation of thoracic diseases. J Thorac Dis. 2013 Aug;5 Suppl 2(Suppl 2):S127-31. doi: 10.3978/j.issn.2072-1439.2013.07.41. PMID 23977433
- [Background] Liu Y, Wong KK, Ko EY, Chen X, Huang J, Tsui SK, Li TC, Chim SS. Systematic Comparison of Bacterial Colonization of Endometrial Tissue and Fluid Samples in Recurrent Miscarriage Patients: Implications for Future Endometrial Microbiome Studies. Clin Chem. 2018 Dec;64(12):1743-1752. doi: 10.1373/clinchem.2018.289306. Epub 2018 Sep 20. PMID 30237148
- [Background] Chan CWH, Leung TF, Choi KC, Tsui SKW, Chan JYW. Effects of gut microbiome and environment on the development of eczema in Chinese infants. Medicine (Baltimore). 2020 May 22;99(21):e20327. doi: 10.1097/MD.0000000000020327. PMID 32481318
- [Background] Wong SH, Yu J. Gut microbiota in colorectal cancer: mechanisms of action and clinical applications. Nat Rev Gastroenterol Hepatol. 2019 Nov;16(11):690-704. doi: 10.1038/s41575-019-0209-8. Epub 2019 Sep 25. PMID 31554963
- [Background] Yu J, Feng Q, Wong SH, Zhang D, Liang QY, Qin Y, Tang L, Zhao H, Stenvang J, Li Y, Wang X, Xu X, Chen N, Wu WK, Al-Aama J, Nielsen HJ, Kiilerich P, Jensen BA, Yau TO, Lan Z, Jia H, Li J, Xiao L, Lam TY, Ng SC, Cheng AS, Wong VW, Chan FK, Xu X, Yang H, Madsen L, Datz C, Tilg H, Wang J, Brunner N, Kristiansen K, Arumugam M, Sung JJ, Wang J. Metagenomic analysis of faecal microbiome as a tool towards targeted non-invasive biomarkers for colorectal cancer. Gut. 2017 Jan;66(1):70-78. doi: 10.1136/gutjnl-2015-309800. Epub 2015 Sep 25. PMID 26408641
- [Background] Ng CF, Chiu PKF, Yee CH, Lau BSY, Leung SCH, Teoh JYC. Effect of androgen deprivation therapy on cardiovascular function in Chinese patients with advanced prostate cancer: a prospective cohort study. Sci Rep. 2020 Oct 22;10(1):18060. doi: 10.1038/s41598-020-75139-w. PMID 33093594
- See also: Hong Kong Cancer Registry. — https://www3.ha.org.hk/cancereg/topten.html
- See also: Globoscan 2018 — https://gco.iarc.fr/today/data/factsheets/cancers/27-Prostate-fact-sheet.pdf
- See also: EAU-EANM-ESTRO-ESUR-SIOG Guidelines on Prostate Cancer 2019 — https://uroweb.org/guideline/prostate-cancer/#6
- See also: 27. NCCN Clinical Practice Guidelines in Oncology - Asia Consensus Statement - version 2.2013. — https://www.nccn.org/professionals/physician_gls/PDF/prostate-asia.pdf